CLINICAL TRIAL: NCT04450706
Title: FORESEE: Functional Precision Oncology for Metastatic Breast Cancer: a Feasibility Trial
Brief Title: Functional Precision Oncology for Metastatic Breast Cancer
Acronym: FORESEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI131027
Record Dates: First submitted 2020-06-22; First posted 2020-06-29 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: HER2-negative Breast Cancer
MeSH Terms: interventions — Precision Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment: all patients (Experimental): Blood will be collected, and a biopsy will be performed prior to starting the first systemic therapy (triple-negative) or first chemotherapy (hormone receptor-positive). If enough tumor is collected, the patient is eligible for the trial. Malignant tissue collected from this biopsy will be used for genomic sequencing and for the development of organoid models for drug screening. Drugs selected for sensitivity testing will be guided by the results of the genome analysis and NCCN guidelines. Following tissue acquisition, the patient will begin therapy as selected by the treating physician. This first-line of on study therapy, either standard-of-care or investigational in the context of another existing active clinical trial, will be defined as the first "uninformed" line of therapy.
  Patient response is tracked for up to two uninformed lines of therapy. The first line of the therapy started after the biopsy will count as the first uniformed line.
  Interventions: Other: Precision Medicine
- Physician Questionnaire (Experimental): The results from the drug screening and mutation testing will be summarized and returned to the treating physician before the assignment of on study, second-line therapy. Before and after returning results, the treating physician will be administered a survey to assess the potential effect that the precision medicine results have on the selection of the following line of therapy. If a patient begins a therapy that was recommended by the precision medicine results, the therapy will be defined as the "informed" line of therapy.
  Interventions: Other: Physican Decision Making

INTERVENTIONS:
Other: Precision Medicine — The tissue from the participant sample will be used for genome sequencing and organoid establishment for drug screening. Both solid tumor genome analysis (commercial and Welm genome) must be performed on tissue from the same biopsy. After the biopsy, the patient will begin uninformed therapy (standard of care or investigational in the context of a separate existing active clinical trial), as selected and directed by the treating physician. Once the results from the genome sequencing and drug screening are available, they will be returned to the treating physician. Upon progression on the uninformed line of therapy, the patient will begin a new therapy as directed by the treating physician. If the patient begins a therapy recommended by the precision oncology results then the next line of therapy will be deemed "informed". While receiving the therapy, response assessments will be conducted until documented radiographic or clinical progression.
  Arms: Treatment: all patients
Other: Physican Decision Making — The results from the drug screening and mutation testing will be summarized and returned to the treating physician before the assignment of on study, second-line therapy. Before and after returning results, the treating physician will be administered a survey to assess the potential effect that the precision medicine results have on the selection of the following line of therapy. If a patient begins a therapy that was recommended by the precision medicine results, the therapy will be defined as the "informed" line of therapy.
  Arms: Physician Questionnaire

SUMMARY:
This is a pilot study to assess the feasibility of comprehensive genomic characterization and drug screening in metastatic breast cancer. The trial will seek to provide personalized genomic and drug sensitivity information to eligible patients with metastatic breast cancer prior to disease progression on standard treatment. The trial will also explore how these results influence physician selection of next-line therapy.

DETAILED DESCRIPTION:
The study will enroll patients with Her2 negative (negative on immunohistochemistry or nonamplified by immunofluorescence in situ hybridization) metastatic breast cancer. Cohorts will enroll according to patient hormone receptor status as hormone receptor-positive or triple-negative. In Part 2, the trial will enroll six patients with triple-negative breast cancer and six patients with ER and/or PR receptor-positive breast cancer. Patients diagnosed with metastatic disease upfront or after a variable interval from completion of definitive therapy for local or locally advanced breast cancer will be eligible.

Patients with triple-negative metastatic breast cancer will be offered to participate in the trial at the time of diagnosis. Patients with hormone receptor-positive disease will be offered the option to participate in the study when they have exhausted endocrine monotherapy or endocrine therapeutic combinatorial options. Blood will be collected, and a biopsy will be performed prior to starting the first systemic therapy (triple-negative) or first chemotherapy (hormone receptor-positive). If enough tumor is collected, the patient will be deemed eligible for the trial. Malignant tissue collected from this biopsy will be used for genomic sequencing and for the development of organoid models for drug screening. Drugs selected for sensitivity testing will be guided by the results of the genome analysis and NCCN guidelines. Following tissue acquisition, the patient will begin therapy as selected by the treating physician. This first-line of on study therapy, either standard-of-care or investigational in the context of another existing active clinical trial, will be defined as the first "uninformed" line of therapy.

The results from the drug screening and mutation testing will be summarized and returned to the treating physicianbefore the assignment of on study, second-line therapy. Before and after returning results, the treating physician will be administered a survey to assess the potential effect that the precision medicine results have on the selection of the following line of therapy. If a patient begins a therapy that was recommended by the precision medicine results, the therapy will be defined as the "informed" line of therapy.

Patient response will be tracked for up to two uninformed lines of therapy. The first line of therapy started after the biopsy will count as the first uniformed line. If a patient does not begin an informed line of therapy after two lines of uninformed therapy they will be taken off study. Response and time of progression will be recorded on both informed and uninformed lines of therapy.

The trial will open to enrollment in two stages. Stage One will enroll three patients to assess preliminary program feasibility and to optimize the genomics pipeline and time frames. After enrollment of the first three patients, enrollment will be put on hold. Upon return of results to the treating physicians, the genomics pipeline and time frames will be evaluated. If necessary, the process will be amended to maximize pipeline efficiency and decrease the interval of time between tumor tissue acquisition and the return of results.

Stage Two will enroll 12 additional patients to further evaluate on a larger scale our functional precision oncology program in metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Her2 negative on immunohistochemistry or nonamplified breast cancer
* Metastatic or recurrent unresectable breast cancer:

  * Patient with triple-negative breast cancer without prior treatment in the metastatic setting.
  * OR
  * Patient with hormone receptor-positive breast cancer that has exhausted or refused all endocrine monotherapy or endocrine therapeutic combinatorial options AND has not yet been treated with chemotherapy in the metastatic settings, but for whom chemotherapy is indicated.
* Willing and capable (per treating investigator's assessment) to undergo baseline tumor collection. Tumor collection may include a solid tumor tissue sample or a fluid sample containing tumor cells.
* Patient can safely undergo tumor collection:

  * The tumor is reasonably accessible to tumor collection;
  * The tumor is amenable to tumor collection, e.g. does not abut neurovascular structures;
  * If the patient receives anticoagulation, anticoagulation can be safely withheld to accommodate for tissue acquisition;
  * The patient does not have a medical condition that would render tumor acquisition a high-risk procedure, (e.g. tumor material acquisition from lung metastases in a patient with emphysema).
* Life expectancy of ≥ 6 months as assessed by the treating investigator.
* ECOG Performance Status ≤ 2.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have estradiol and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* At least one lesion (measurable or non-measurable) that can be accurately assessed at baseline and is suitable for repeated assessment by computed tomography (CT), magnetic resonance imaging (MRI), plain X-ray, or physical examination.

Exclusion Criteria:

* Diagnosis of any other malignancy with a life expectancy of < 5 years.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (> New York Heart Association Classification Class IIB) or a serious cardiac arrhythmia requiring medication.
  * Renal or liver disease that prohibits the patient from receiving at least single-agent full recommended dose chemotherapy.
* The patient cannot safely undergo tumor collection for reasons including but not limited to:

  * Tumor is inaccessible;
  * The patient requires anticoagulation which cannot be withheld;
  * The patient has bleeding diathesis;
  * Any other reason that would render tumor tissue acquisition a high-risk procedure.
* Patient cannot or is unwilling to receive chemotherapy
* Known brain metastases or cranial epidural disease. Note: Brain metastases or cranial epidural disease adequately treated with radiotherapy and/or surgery and stable for at least 4 weeks before Step 1 Registration for study will be allowed on trial. Subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the Step 1 Registration for study.
* Patient's only site amenable to tumor collection to generate organoids is hepatic metastases.

Physician Inclusion Criteria

* Physician is the treating medical oncologist for a patient who meets all of the inclusion criteria and none of the exclusion criteria.
* Willing and able to answer the physician questionnaires at the protocol required time points.
* Willing and able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Organoid Development and Tumor Material Testing Patient Eligibility

* Patient continues to meet step 1 registration criteria.
* Successful acquisition of a solid tumor biopsy sample containing ≥ 20% tumor content, or malignant fluid sample (e.g. pleural or pericardial effusion or ascites) confirmed to contain malignant cells.
* Sufficient material for Tempus commercial genomics testing and Welm lab genomics from the tumor collection; or sufficient archival tissue for Tempus and Welm lab genomics; or blood sample as allowed for liquid biopsy commercial assay.
* Sample from tumor collection is the type of sample that is feasible for organoid development as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Number of cases where clinically actionable outcomes were identified by the use of organoids and drug screening (functional precision oncology). | 12 weeks
  Determine the feasibility of comprehensive genomic characterization and drug screening for metastatic breast cancer in a clinically relevant time frame.

SECONDARY OUTCOMES:
The time from patient sample collection to return of genomic characterization results. | up to 2 years
  Time required to return genomic characterization and drug screening results to treating physicians
The time from patient sample collection to return of drug screening results. | up to 2 years
  Time required to return genomic characterization and drug screening results to treating physicians
Performance: comparison between the number of clinically actionable outcomes identified by our functional genomic characterization and commercially available assays | up to 2 years
  assess the performance and concordance of our integrated functional genomic assays (drug screen with or without genomic characterization) against commercially available assays.
Concordance: To assess the frequency with which our functional precision oncology testing identifies the same therapeutic vulnerabilities identified by commercial (gold standard) testing. | up to 2 years
  assess the performance and concordance of our integrated functional genomic assays (drug screen with or without genomic characterization) against commercially available assays.

CONTACTS AND LOCATIONS:
Overall Officials: Saundra Buys, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No